CLINICAL TRIAL: NCT06548113
Title: Investigation of Sensory Synchronized Human Brain Imaging and Neuromodulation
Brief Title: Sensory Synchronized Imaging and Neuromodulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: MHBC-011-24F; 76106 (Other: VA Palo Alto Health Care System)
Record Dates: First submitted 2024-08-01; First posted 2024-08-12 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard TMS (Active Comparator): A series of standard TMS protocols will be delivered to determine target engagement compared to seTMS. TMS will be delivered using neuro-navigation based on participant's own MRI images. Intensity will be set to 120% of the participant's motor threshold. Participants will be monitored during the session for adverse events and/or side effects.
  Interventions: Device: TMS
- Sensory-entrained TMS (seTMS) (Active Comparator): Sensory entrained TMS (seTMS) is a combination of music and TMS to align brain oscillations and enhance the effects of TMS. seTMS will be delivered to determine target engagement to noninvasive seTMS brain stimulation compared to standard TMS. TMS will be delivered using neuro-navigation based on participant's own MRI images. Intensity will be set to 120% of the participant's motor threshold. Participants will be monitored during the session for adverse events and/or side effects.
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS — transcranial magnetic brain stimulation

SUMMARY:
The purpose of this research study is to better understand the relationship between the type of brain stimulation used and how it changes brain activity in adult military Veterans. The goal is to use this understanding to develop new, personalized brain stimulation. The investigators evaluate brain changes from different types of transcranial magnetic brain stimulation (TMS).

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages 18 years and up
* English speaking
* Military Veterans

Exclusion Criteria:

* Those with a contraindication for MRIs (e.g. implanted metal)
* History of head trauma with loss of consciousness
* History of seizures or on medications that substantially reduce seizure threshold
* Neurological or uncontrolled medical disease
* Active substance abuse
* Currently pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2029-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Transcranial Magnetic Stimulation (TMS) / Electroencephalography (EEG) change | 45 minutes
  Change in the TMS-EEG measure will be assessed before, during, and after each TMS session. Specifically, the difference in size of the evoked response after a single TMS pulse in the frontoparietal region will be quantified in microVolts and compared between standard TMS and sensory-entrained TMS (se-TMS).

CONTACTS AND LOCATIONS:
Overall Officials: Jessica M Ross, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No